CLINICAL TRIAL: NCT02086019
Title: A Prospective Randomised Controlled Trial
Brief Title: Revascularisation or Medical Therapy in Elderly Patients With Acute Anginal Syndromes
Acronym: RINCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Principal Investigator, Adam de Belder, Consultant Cardiologist, Brighton and Sussex University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN-AdB-RINCAL-2013
Record Dates: First submitted 2014-03-04; First posted 2014-03-13 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Acute Coronary Syndromes
Keywords: Revascularisation, octogenarian,acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Heparin, Low-Molecular-Weight; Aspirin; Clopidogrel; Adrenergic beta-Antagonists; Bisoprolol; Angiotensin-Converting Enzyme Inhibitors; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative Arm- Medical therapy (Other): Medical therapy
  Interventions: Drug: Conservative Arm
- Invasive Arm-angiogram with PCI or CABG (Other): same medical drug therapy as conservative arm, and angiogram with PCI (percutaneous coronary intervention) or CABG (coronary artery bypass grafting) revascularisation if appropriate
  Interventions: Procedure: Invasive Arm

INTERVENTIONS:
Drug: Conservative Arm — crossover to angiogram only if predefined criteria met
  Other Names: low molecular weight heparin,; aspirin,; clopidogrel,; beta blocker (Bisoprolol or equivalent); ACE inhibitor (Ramipril or equivalent)
  Arms: Conservative Arm- Medical therapy
Procedure: Invasive Arm — angiogram with PCI or CABG revascularisation if appropriate
  Arms: Invasive Arm-angiogram with PCI or CABG

SUMMARY:
For octogenarian patients with NSTEMI (non-ST segment elevation myocardial infarction) an invasive-guided strategy will prove superior to a conservative strategy with respect to a combined endpoint of all cause mortality and non-fatal myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* AGE>80 Non-STEMI - characteristic chest pain accompanied by
* Typical ischaemic ECG changes
* A troponin rise

Suitable for conservative or invasive strategy

Exclusion Criteria:

* Lack of suitability for whatever clinical reason to be randomised eg dementia, co-morbidity
* Acute STEMI
* Cardiogenic shock
* Platelet count =50 x 109/mm3
* Patient life expectancy < 1 year
* Known allergies to clopidogrel, aspirin, heparin, stainless steel, IV contrast or stent drug elutant
* Recent major GI haemorrhage (within 3 months)
* Any previous cerebral bleeding episode
* Participation in another investigational drug or device study
* Patient unable to give consent
* Clinical decision precluding the use of stents

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-05-01; Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Death | 1 year
  The cause of death will be adjudicated as being due to cardiovascular causes, non cardiovascular causes, or undetermined causes.
  * Cardiovascular Death includes sudden cardiac death, death due to acute myocardial infarction, death due to heart failure or cardiogenic shock, death due to stroke or death due to other cardiovascular causes
  * Non-Cardiovascular Death is defined as any death not covered by cardiac death or vascular death.
  * Undetermined cause of death refers to a death not attributable to one of the above categories of cardiovascular death or to a non-cardiovascular cause.
  N.B For this trial all deaths with undetermined causes will be included in the cardiovascular category.
non-fatal myocardial infarction | 1 year
  The ESC/ACC (European Society of Cardiology and the American College of Cardiology) definition of myocardial infarction will be applied, including the special circumstances of same admission myocardial re-infarction, or myocardial infarction peri-PCI.

SECONDARY OUTCOMES:
Unplanned revascularisation | 1 years
  Shall be deemed to have occurred at follow-up if any coronary vessel requires or undergoes attempted repeat revascularisation with either balloon angioplasty, stenting, or coronary artery bypass grafting.
Permanent Stroke | 1 year
  A stroke is a loss of neurological function caused by an ischemic or hemorrhagic event with residual symptoms at least 24 hours after onset or leading to death
Major bleeding | 1 year
  BARC (Bleeding Academic Research Consortium) definition
Deterioration of renal function during hospital admission | During index admission
  Worsening renal function is an absolute increase in serum creatinine of ≥ 0.3mg/dl (26.5 umol/l) at any time during hospitalization compared to the valve obtained at admission
Angina symptoms (3 months; 1yr) | 3 months and 1 year
  CCS (Canadian Cardiovascular Society Classification of angina) grading of angina
Stent thrombosis | 1 year
  ARC definition of stent Thrombosis
All cause mortality | 2,3 and 4 year
  Cardiac and non cardiac mortality
Hospital readmission for ACS/STEMI | At 3, 6 and 12 months and at 2,3 and 4 years
  ESC/ACC definition ACS/STEMI (Acute coronary syndrome/ST-segment elevation myocardial infarction)
In-hospital major complications | At 3, 6 and 12 months and at 2,3 and 4
  In hospital major complications defined as death, myocardial infarction, stent thrombosis, target restenosis, repeat target- and non-target vessel-related percutaneous coronary intervention, target lesion revascularization, coronary artery bypass surgery and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Sussex County Hospital, Brighton, United Kingdom